CLINICAL TRIAL: NCT00222469
Title: A Phase II Trial of Bevacizumab Plus Gemcitabine™ and Oxaliplatin™ as First Line Therapy in Metastatic or Locally Advanced (Unresectable) Pancreatic Cancer
Brief Title: Combination Chemotherapy for 1st Line Treatment of Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Genentech, Inc. (Industry); Sanofi (Industry); M.D. Anderson Cancer Center (Other)
Responsible Party: Mehrdad Jafari, MD, University of Oklahoma Dept. of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2004-0652
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; unresectable pancreatic cancer; metastatic pancreatic cancer; bevacizumab; oxaliplatin; gemcitabine; 1st line treatment; first line treatment; locally advanced (unresectable) pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Oxaliplatin

ARMS (1):
- 1 (Experimental): 3-agent treatment group
  Interventions: Drug: bevacizumab; Drug: gemcitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: bevacizumab — 10mg/kg IV on Day 1 Q 2 weeks
Drug: gemcitabine — 1000mg/m2 as fixed-rate infusion at 10mg/m2/min on Day 1 and Q 2 weeks.
Drug: oxaliplatin — 100mg/m2 on Day 2 and Q 2 weeks.

SUMMARY:
The purpose of this study is to find out if giving patients bevacizumab along with the chemotherapy drugs oxaliplatin and gemcitabine will improve overall survival.

In addition, the study will find out what side effects patients may have by taking bevacizumab, oxaliplatin, and gemcitabine together.

DETAILED DESCRIPTION:
Design:

* A phase II single arm study. All patients receive bevacizumab 10mg/kg and gemcitabine 1000mg/m2 on day 1 followed by oxaliplatin 100mg/m2 on day 2 of a 14 day cycle.

Purpose:

* The purpose of this study is to find out if giving patients bevacizumab, along with the chemotherapy drugs oxaliplatin and gemcitabine, will improve overall survival. In addition, the study will find out what side effects patients may have by taking bevacizumab, oxaliplatin and gemcitabine together.

Enrollment:

* Approximately 30 patients will be enrolled to the study between the University of Oklahoma and M.D. Anderson Cancer Center.

Duration:

* The study will be conducted over approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years old
* ECOG performance status 0-2.
* Patients with metastatic or unresectable locally advanced adenocarcinoma of the pancreas.
* Patients who have recurrent disease post pancreaticoduodenectomy no earlier than 6 months after resection. Patients with recurrent disease who had completed adjuvant therapy in the form of radiation with or without radiosensitizing 5-fluorouracil (5-FU) 6 months prior to recurrence may be included.
* Signed informed consent/authorization is obtained prior to conducting any study specific screening procedures.
* No prior chemotherapy for advanced pancreatic cancer
* Patient must have measurable disease
* Use of effective means of contraception (men and women) in subjects of child-bearing potential
* Obstructive jaundice must be relieved before inclusion
* Adequate hepatic, renal, and bone marrow function: leukocytes >= 3,000/uL, absolute neutrophil count >= 1,500/uL, platelets >= 100,000/uL, total bilirubin < = 1.5 X institutional upper limits of normal (ULN), AST (SGOT)/ALT (SGPT) <= 2.5 X institutional ULN, creatinine <= 1.5 mg/dL

Exclusion Criteria:

* Previous chemotherapy for pancreatic cancer.
* Patients who have recurrent disease within 6 months after pancreaticoduodenectomy or had received adjuvant therapy within 6 months of disease recurrence.
* Uncontrolled intercurrent illness including:

  * Active infection
  * Cardiovascular: New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months, blood pressure > 150/100 mmHg
  * Clinically significant peripheral vascular disease
  * History of stroke within previous 6 months
  * Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0
* Urine protein:creatinine ratio > 1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events. A computed tomography (CT) scan of the brain is not needed for eligibility and will be done only if the patient presents with symptoms suggestive of brain metastases.
* Patients may not be receiving any other investigational agents, or have participated in any investigational drug study within 28 days preceding start of study treatment.
* The teratogenic potential of this combination is currently unknown. Women who are pregnant or lactating are excluded.
* History of any other malignancy in the last 5 years, except patients with a prior history of in situ cancer or basal or squamous cell skin cancer.
* Peripheral neuropathy > grade 1
* Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To determine the overall survival (OS) rate at 1 year in this patient population, treated with the combination therapy of bevacizumab plus gemcitabine and oxaliplatin | One year

SECONDARY OUTCOMES:
To determine the objective tumor response rate in this patient population. To determine time to progression (TTP) and progression free survival (PFS) in this patient population | One year
To determine the tolerability and toxicity profile of this regimen in this patient population | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Jafari, MD, PhD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Oklahoma, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas